CLINICAL TRIAL: NCT02374437
Title: Pharmacokinetics of Single and Multiple Escalating Doses of Aramchol and Food Effect in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Aramchol004
Record Dates: First submitted 2015-01-18; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — aramchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- PART A (single dose)-200 mg (Active Comparator): 200 mg ARAMCHOL
  Interventions: Drug: Aramchol
- PART A (single dose)-400 mg (Active Comparator): 400 mg ARAMCHOL
  Interventions: Drug: Aramchol
- Part B ( food effect)- -Fasting (Active Comparator): 600 mg Aramchol tablets under fasting conditions (fasting for at least 10 hours before and 4 hours after dosing)
  Interventions: Drug: Aramchol
- Part B ( food effect)- -Fed (Active Comparator): 600 mg Aramchol tablets under fed conditions (fasting for at least 10 hours before dosing, consumption of a high calorie high fat meal within 30 minutes prior to drug administration and no food for additional 4 hours after dosing)
  Interventions: Drug: Aramchol
- Part C ( multiple doses)- 200 mg (Active Comparator): 200 mg Aramchol tablets for ten consecutive days.
  Interventions: Drug: Aramchol
- Part C ( multiple doses)- 400 mg (Active Comparator): 400 mg Aramchol tablets for ten consecutive days.
  Interventions: Drug: Aramchol
- Part C ( multiple doses)- 600 mg (Active Comparator): 600 mg Aramchol tablets for ten consecutive days.
  Interventions: Drug: Aramchol
- Part C ( multiple doses)- Placebo (Placebo Comparator): Placebo tablets for ten consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aramchol — PART A: Subjects will receive single dose of 200 or 400 mg Aramchol PART B: Subjects will receive single dose of 600 mg Aramchol under fasting or fed conditions ( following a crossover between the groups) PART C: subjects will be equally randomized to receive either 200 mg, 400 mg, 600 mg or placebo tablets for ten consecutive days.
  Arms: PART A (single dose)-200 mg; PART A (single dose)-400 mg; Part B ( food effect)- -Fasting; Part B ( food effect)- -Fed; Part C ( multiple doses)- 200 mg; Part C ( multiple doses)- 400 mg; Part C ( multiple doses)- 600 mg
Drug: Placebo — PART C: subjects will be equally randomized to receive either 200 mg, 400 mg, 600 mg or placebo tablets for ten consecutive days.
  Arms: Part C ( multiple doses)- Placebo

SUMMARY:
This is a single-site, randomized, partly double-blind, placebo-controlled study of Aramchol in sixty six (66) healthy male volunteers.

In each part of the study subjects will be enrolled in the study within 28 days before drug administration(s).

The study will consist of three parts and the subjects will be assigned to three Parts.

DETAILED DESCRIPTION:
This is a single-site, randomized, partly double-blind, placebo-controlled study of Aramchol in sixty six (66) healthy male volunteers.

In each part of the study subjects will be enrolled in the study within 28 days before drug administration(s).

The study will consist of three parts and the subjects will be assigned to three Parts as follows:

Part A - single escalating doses:

The purpose of this part is to evaluate the pharmacokinetics, safety and tolerability of Aramchol tablets at single doses of either 200 mg or 400 mg.

Twelve (12) subjects will be randomized to receive , following an overnight 10 hours fast, a single dose of either:

* Administration A: 1×200 mg Aramchol tablet (6 subjects)
* Administration B: 1×400 mg Aramchol tablet (6 subjects) Subjects will be admitted to the Clinical Research Center (CRC) in the evening before study drug administration (Day 0) and will remain in-house for 36 hours after dosing. Blood samples for Aramchol concentrations will be drawn for 36 hours at designated time points as described below. Additional ambulatory samples will be collected at 48, 72, 96 and 144 hours post-dose. Subjects will be continuously monitored for safety.

An End-of Study/Safety Follow-up visit will take place on the last PK sampling day, i.e. 144 hours post-dose.

Part B - food effect:

The purpose of this part is to evaluate the effect of high fat high calorie meal on the pharmacokinetics of a single dose of Aramchol and to assess the safety and tolerability of a single 600 mg dose.

This part is designed as a randomized, two period crossover food-effect study.

Eighteen (18) subjects will be randomized to receive one of two administration sequences (C-D or D-C) as follows:

* Administration C: 1×200 mg +1×400 mg Aramchol tablets under fasting conditions (fasting for at least 10 hours before and 4 hours after dosing)
* Administration D: 1×200 mg +1×400 mg Aramchol tablets under fed conditions (fasting for at least 10 hours before dosing, consumption of a high calorie high fat meal within 30 minutes prior to drug administration and no food for additional 4 hours after dosing) In each period of this part, subjects will be admitted to the Clinical Research Center (CRC) in the evening before study drug administration (Day 0) and will remain in-house for 36 hours after dosing. Blood for Aramchol concentrations will be drawn for 36 hours at designated time points as described below. Additional ambulatory samples will be collected at 48, 72, 96 and 144 hours post-dose. Subjects will be continuously monitored for safety.

There will be a wash-out period of at least 14 days between each dosing session.

An End-of Study/Safety Follow-up visit will take place on the last PK sampling day of the second dosing period, i.e. 144 hours after second dose.

The PK profile of subjects who received administration C (i.e. 600 mg Aramchol tablet under fasting conditions) will be compared with that of subjects who received 200 and 400 mg Aramchol tablet under fasting conditions in Part A.

Part C - multiple doses:

The purpose of this part is to evaluate the pharmacokinetics, safety and tolerability of Aramchol tablets at multiple administrations of 3 different doses.

This part is designed as a randomized, double blind, double-dummy, placebo-controlled multiple-dose study.

Thirty six (36) subjects will participate in this part and will be equally randomized to receive either 200 mg, 400 mg, 600 mg or placebo tablets for ten consecutive days. Drug administration will be preceded by a light breakfast consumed within 1 hour prior to dosing (the composition of which is described in Appendix III). All drugs will be administered by the study staff except Dose No. 6 which the subjects will take at home.

In order to maintain blinding, all subjects will receive two tablets on each dosing, according to the following administrations:

* Administration E: 1×200 mg Aramchol tablet + 1×400 mg Placebo tablet
* Administration F: 1×200 mg Placebo tablet + 1×400 mg Aramchol tablet
* Administration G : 1×200 mg Aramchol tablet + 1×400 mg Aramchol tablet
* Administration H: 1×200 mg Placebo tablet + 1×400 mg Placebo tablet

Treatment assignment will be as follows:

Subjects will be admitted to the Clinical Research Center (CRC) in the evening before the first study drug administration (Day 0) and will remain in-house for 24 and 36 hours after first (Day 1) and last (Day 10) doses, respectively. PK blood samples will be drawn on Day 1 for 24 hours at designated time points as described below. Additionally, ambulatory pre-dose (trough) samples will be drawn before dosing on Days 2, 3, 4, 5, 7, 8, and 9. On Day 10 blood samples will be collected for 36 hours at designated time points as described below and during additional ambulatory visits at 48, 96, 120, 144, 168 and 192 hours post-dose.

Subjects will be continuously monitored for safety. An End-of Study/Safety Follow-up visit will take place on the last PK sampling day of the study, i.e. 144 hours (for Parts A and B) and 192 hours (for Part C) after the last dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, males subjects between 18-50 years (inclusive)
2. 21.0<BMI< 29.9kg/m2
3. Non-smoking (by declaration) for a period of at least 3 months before screening visit.
4. Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
5. No significant abnormalities in ECG (e.g. prolonged QTC, prolonged PR interval) done at screening and on Days (0) before dosing session.
6. No clinically significant abnormalities in hematology, blood chemistry, or urinalysis lab tests at screening.
7. No known history of alcohol or drug abuse. Subjects with negative urinary drugs of abuse screen determined on Day (0) before dosing session(s)
8. Negative HIV, hepatitis B or hepatitis C serology tests as evaluated at screening.
9. Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
10. Subjects must agree to use adequate birth control measures (condom in combination with a spermicidal gel or foam) during the study and up to 15 days after the last study drug administration.
11. Subjects must satisfy a medical examiner about their fitness to participate in the study.
12. Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Documented history or on-going symptoms of any gastrointestinal disorder involving motility, gastric acid or gastric emptying or malabsorption, including but not limited to, peptic ulcer disease, gastroesophageal reflux, dyspepsia, gastroparesis, chronic diarrhea, chronic constipation, gall bladder disease, pancreatitis, lactose intolerance and celiac disease.
2. History of esophageal, gastric, biliary, or intestinal surgery (excluding herniotomy and appendectomy which are not related to gastrointestinal disorders).
3. Known history of significant medical disorder, which in the investigator's judgment contraindicates administration of the study medications.
4. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit.
5. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol or ibuprofen for symptomatic relief of pain is allowed until 24 hours prior to the study drug administration.
6. Subjects who have taken anticholinergic or other drugs known to affect gastrointestinal motility within 7 days prior to the first dosing
7. Treatment with any drugs with known hepatic enzyme-inducing or inhibiting agents (such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc.) within 30 days prior to dosing.
8. Known hypersensitivity and/or allergy to any drugs.
9. Adherence (for whatever reason) to an abnormal diet during the 4 weeks prior to the study, or subjects with recent significant change in body weight
10. Any acute illness (e.g. acute infection) within 48 hours prior to the first study drug administration, which is considered of significance by the Principal Investigator.
11. Participation in another clinical trial with drugs, received within 3 months prior to dosing (calculated from the previous study's last dosing date).
12. Subjects who donated blood in the three months or received blood or plasma derivatives in the six months preceding study drug administration.
13. Subjects with inability to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).
14. Inability to fast or consume the food provided in the study (including any known food allergies or food restrictions).
15. Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose. Part C:Dosing days 1-10
Area under the plasma concentration time curve (AUC) | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose. Part C:Dosing days 1-10
Maximum plasma concentration (Cmax) | Part B: For each treatment period: Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72(±60 min), 96(±60 min), 144 (±60 min) hours post dose.
Area under the plasma concentration time curve (AUC) | Part B: For each treatment period: Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72(±60 min), 96(±60 min), 144 (±60 min) hours post dose.
Maximum plasma concentration (Cmax) | Part C: day 1 and day 10
Area under the plasma concentration time curve (AUC) | Part C: day 1 and day 10

SECONDARY OUTCOMES:
Adverse event (AE) profile | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose. Part C:Dosing days 1-10
  Adverse event records in patients file
Adverse event (AE) profile | Part B: For each treatment period: Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72(±60 min), 96(±60 min), 144 (±60 min) hours post dose.
  Adverse event records in patients file
Adverse event (AE) profile | Part C:Dosing days 1 and 2: pre-dose (within 60 min before first dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18 and 24 (before second dosing) hours after drug administration+ day 3-10
  Adverse event records in patients file
Clinical laboratory safety tests | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose. Part C:Dosing days 1-10
  blood test
Clinical laboratory safety tests | Part B: For each treatment period: Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72(±60 min), 96(±60 min), 144 (±60 min) hours post dose.
  blood test
Clinical laboratory safety tests | Part C:Dosing days 1 and 2: pre-dose (within 60 min before first dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18 and 24 (before second dosing) hours after drug administration+ day 3-10
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: Maya Halpern, MD, Study Director — GALMED PHARMCEUTICALS